CLINICAL TRIAL: NCT01698281
Title: A Randomized Phase 2 Trial of AEZS-108 in Chemotherapy Refractory Triple Negative, LHRH-positive Metastatic Breast Cancer.
Brief Title: Phase 2 Trial of AEZS-108 in Chemotherapy Refractory in Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEZS-108-049
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2013-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — LHRH, lysine(6)-doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: AEZS-108 (Experimental): Intervention: AEZS-108 (267 mg/m^2, 2-hour IV infusion every Day 1 of a 21-day (3-week) cycle). Recommended prophylactic anti-emetic for AEZS-108: 8 mg dexamethasone
  Interventions: Drug: AEZS-108; Drug: Dexamethasone
- Arm B: Standard (SCCC) (Active Comparator): commercially available standard single agent cytotoxic chemotherapy (SSCC): - doses below the recommended package insert at the discretion of treating oncologist;
  - on a 21-day cycle (although weekly administration is allowed; note: pegylated liposomal doxorubicin will be administered on a 28-day cycle).
  Interventions: Drug: SCCC

INTERVENTIONS:
Drug: AEZS-108 — AEZS-108 (267 mg/m2, 2-hour IV infusion every Day 1 of a 21-day (3-week) cycle. Allowed delay of re-treatment: up to 2 weeks.
  Dose reduction: to 210 mg/m2 and 160 mg/m2, if dose limiting toxicity.
  Other Names: Zoptarelin doxorubicin
  Arms: Arm A: AEZS-108
Drug: SCCC — commercially available SSCC (doses below the recommended package insert at the discretion of treating oncologist), on a 21-day cycle (although weekly administration is allowed; note: pegylated liposomal doxorubicin will be administered on a 28-day cycle).
  Drugs considered acceptable as SSCC: paclitaxel; nab-paclitaxel; eribulin; pegylated liposomal doxorubicin (PLD); vinorelbine; gemcitabine; capecitabine.
  Related to PLD: Per notification from EMA (dated 22-Nov-2011) "no new patients should be started on treatment with Caelyx until further notice." Accordingly, this drug may be selected as SSCC treatment option only after such written notice is available.
  Other Names: Standard single agent cytotoxic chemotherapy
  Arms: Arm B: Standard (SCCC)
Drug: Dexamethasone — Recommended prophylactic anti-emetic for AEZS-108: 8 mg dexamethasone.
  Arms: Arm A: AEZS-108

SUMMARY:
This is a therapeutic exploratory Phase 2 study evaluating AEZS-108 compared to standard single agent cytotoxic chemotherapy (SSCC) as measured by the median time of progression-free survival (PFS) in patients with chemotherapy refractory triple negative (ER/PR/HER2-negative) LHRH-R positive metastatic breast cancer.

DETAILED DESCRIPTION:
The study will be conducted as an open-label randomized two-arm multicenter Phase II study. Patients will be randomized in a 1:1 ratio into one of the two treatment arms within each stratum: AEZS-108 (267 mg/m2 every 21 calendar days) (Arm A) OR SSCC (Arm B) at discretion of treating oncologist cycled every 21 calendar days.

Stratified randomization will be used with number of prior lines of therapies (1-2 versus >2). Tumor assessment will be repeated every 2 cycles. At the time of disease progression, Arm B patients may be crossed over to AEZS-108 as long as none of the exclusion criteria for study entry apply. Particularly, LVEF ≥50% is required, and patients failing on liposomal doxorubicin cannot be crossed over to AEZS-108.

Analysis of the main study endpoint, PFS, will follow a group sequential design with one interim and one final analysis utilizing the O'Brien-Fleming stopping boundaries procedure. The study will be terminated for futility if the lower bound is crossed and for superiority if the upper bound is crossed. The sponsor may also terminate the study for futility based on other considerations such as safety.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age
2. Histologically documented breast cancer (either primary or metastatic site) that is (i) ER-negative (0), (ii) PR-negative (0), and (iii) HER2-negative, defined by IHC (immunohistochemistry; IHC 0/1, non-overexpressing) or FISH (fluorescence in situ hybridization; FISH negative) or CISH (chromogen in situ hybridization; CISH negative).
3. Expression of LHRH receptor confirmed by IHC on archival (or current biopsy of breast tumor or metastatic site) breast cancer tissue
4. Progressive disease after failure of 1 to 3 prior chemotherapy regimens for recurrent or metastatic (Stage IV) disease (prior adjuvant/neoadjuvant therapy is allowed)
5. Measurable disease by RECIST 1.1 criteria; at least one target lesion that has not been previously irradiated.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status > 2
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or recent myocardial infarction (within 6 months of enrollment)
3. Leptomeningeal disease or brain metastases requiring steroids or other therapeutic intervention
4. Left ventricular ejection fraction (LVEF) < 50 %, determined by echocardiogram or MUGA scan
5. Compromised organ or marrow function as evidenced by any of the following:

   * thrombocyte count: < 100x109/L
   * absolute neutrophil count (ANC): < 1.5x109/L
   * hemoglobin: < 6.0 mmol/L (< 9 g/100 mL)
   * AS(A)T, AL(A)T: > 2.5 times upper limit of normal range (ULN) (> 5x ULN if clearly related to liver metastases)
   * bilirubin: > 1.5 mg/dL
   * creatinine: > 1.5 mg/dL or creatinine clearance < 40 mL/min.
6. Systemic anticancer therapy or radiotherapy within 21 calendar days of the first dose of study drug*)

   * also excluded are patients with anticipated ongoing concomitant anticancer therapy during the study
7. Prior exposure to anthracyclines or anthracenediones for the treatment of metastatic breast cancer including liposomal doxorubicin (Doxil), doxorubicin, daunorubicin, or mitoxantrone
8. Prior adjuvant anthracyclines with a cumulative anthracycline dose ≥ 300 mg/m2
9. Ongoing therapeutic anticoagulation
10. Patients who are not surgically sterile or post-menopausal must agree to use for the duration of the study reliable methods of birth control defined as:

    * complete abstinence
    * any intrauterine device (IUD) with published data showing that the lowest expected failure rate is < 1 % per year, or
    * any other methods with published data showing that the lowest expected failure rate is less than 1 % per year
11. Investigational therapy within 30 calendar days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of AEZS-108 compared to SSCC as measured by the median time of progression-free survival (PFS). | Up to two years
  PFS is defined as the time elapsed from randomization to the date of documented progression or death, whichever comes first. For surviving patients without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.

SECONDARY OUTCOMES:
Efficacy of AEZS-108: overall response | Up to two years
  Overall response per RECIST 1.1 (i.e. complete response (CR) + partial response (PR).
Efficacy of AEZS-108: clinical benefit | up to 2 years
  Overall clinical benefit = complete response (CR) + partial response (PR) + stable disease (SD)
Efficacy of AEZS-108: duration of response | up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
Efficacy of AEZS-108: time to progression (TTP) | up to 2 years
  TTP is defined as the time elapsed from randomization to the earliest date of documented disease progression. For surviving patients without progression of breast cancer who begin alternative treatment, TTP will be censored at the last date of documented progression-free status prior to starting alternative treatment. This is expected to be negligible and, if the actual data suggest otherwise, competing risk methods will be used instead of Kaplan-Meier estimates. Similarly, losses to follow up will be censored at the last date of documented progression free status.
Efficacy of AEZS-108: overall survival | up to 2 years
  Overall survival (OS) is defined as the elapsed time from start of therapy to death from any cause. For surviving patients, follow-up will be censored at the date of last contact.
Toxicity of AEZS-108 in this patient population | up to 2 years
  All patients will be evaluable for toxicity from the time of their first treatment with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J. Montero, MD, Principal Investigator — University of Miami
Locations (3):
- University of Miami, Miami, Florida, United States
- Germany (2):
  - Universitäts-Frauenklinik, Göttingen
  - Klinik für Frauenheilkunde und Geburtshilfe, Regensburg